CLINICAL TRIAL: NCT02058654
Title: A Randomised, Double-blind, Study to Investigate the Effects of Creatine Supplementation on Muscle Energetics and Cognitive Function in Young Healthy Male Athletes and an Ageing Population Using Phosphorus-31 Magnetic Resonance Spectroscopy (31P MRS) and Functional Magnetic Resonance Imaging (fMRI)
Brief Title: A Clinical Study to Investigate the Effects of Creatine Supplementation on Muscle Energetics and Cognitive Function in Young Healthy Male Athletes and an Ageing Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 201131; RH02061 (Other: GSK)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Nutritional Status
Keywords: Creatine; Functional magnetic resonance imaging (fMRI); Phosphorus-31 magnetic resonance spectroscopy (31P-MRS)
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creatine Group (Experimental): Whey protein (30 g) and creatine supplement (5 g) shaken with 250-300 ml water in a blender bottle, and the full shake to be taken twice a day for 14 days.
  Interventions: Drug: Creatine
- Placebo Group (Placebo Comparator): Whey protein (30 g) and bulking agent powder (5 g) shaken with 250-300 ml water in a blender bottle, and the full shake to be taken twice a day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creatine — Creatine powder (5 g)
  Arms: Creatine Group
Drug: Placebo — Bulking agent powder (5 g)
  Arms: Placebo Group

SUMMARY:
This study will examine the impact of creatine supplementation on muscle function and cognitive performance in young and older subjects.

DETAILED DESCRIPTION:
This is a randomised, double-blind study of the effects of creatine supplementation on muscle energetics and cognitive function, using 31P-MRS and fMRI. 31P-MRS data will be acquired continuously during exercise phase and in the post-exercise metabolic recovery phase. Participants will undergo a fMRI scan of the brain to record changes in the blood oxygen level dependent (BOLD) signal during a series of cognitive tests. In addition, participants will undergo a resting state BOLD scan and a structural MRI scan for localization of brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer: Group 1: male; Group 2: male or female.
* Aged 18-35 years (Group 1), or 50-70 years (Group 2).
* Dietary protein intake at or near the current recommended daily amount (0.75 to 0.85 g protein/kg/day).
* Participation in regular physical activity (aerobic and resistance training) 2-3 times a week for at least 6 months before the study starts (Group 1 only).
* Willingness to maintain a stable lifestyle throughout the study.

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory, neurological, or renal function, diabetes mellitus, cardiovascular disease, coagulation disorder, autoimmune disease, phenylketonuria, hyperlipidaemia, or history of any psychotic mental illness.
* Any impairment affecting mobility and muscle metabolism of the lower limbs (such as arthritis).
* Surgery (eg stomach bypass) or medical condition that might affect absorption of supplements.
* Inability to complete the structured exercise program.
* Blood pressure and heart rate in seated position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 35-100 beats/min (Group 1) or 40-100 beats/min (Group 2).
* Metal implants that may affect the MRI scan, eg gold tooth or other metal dental devices (normal dental fillings are allowed), pacemaker, mechanical heart valve, replacement joint, shrapnel. If any metal in the body is identified, the investigators will make a decision, as to whether the subject should participate in the study.
* History of claustrophobia or subject feels unable to lie still on their back for a period of 90 mins in the MRI scanner, or subject unable to perform the required muscle exercise in the MRI scanner.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-24 (Actual)

PRIMARY OUTCOMES:
PCr Concentration (at rest) | Baseline to Day 3, 7 and 14
  Change in PCr concentration (at rest), as measured by 31P- MRS on the calf. Static MRS will be acquired at rest up to 2 min.

SECONDARY OUTCOMES:
PCr concentration during recovery | Baseline to Day 3, 7, and 14
  Change in PCr concentration (during recovery) as measured by 31P- MRS on the calf. Dynamic MRS will be acquired with the patient at rest for up to 20 min.
Change in PCr from rest to recovery | Baseline to Day 3, 7, and 14
  Change in PCr concentration (from rest to recovery) as measured by 31P- MRS on the calf.
PCr recovery rate (PCr(T1/2)) | Baseline to Day 3, 7 and 14
  Measured by 31P-MRS on the leg
ADP recovery rate (ADP (T1/2)) | Baseline to Day 3, 7 and 14
  Measured by 31P-MRS on the leg
pH at the end of pedal test, or at the time of voluntary cessation (Post-pedal test pH) | Baseline to Day 3, 7 and 14
  Measured by 31P-MRS on the leg
Lowest pH measured during pedal test or recovery (Minimum pH) | Baseline to Day 3, 7 and 14
  Measured by 31P-MRS on the leg
BOLD signal in the brain | Baseline to Day 14
  Change in BOLD signal, as measured by an fMRI scan of the brain. Data may be examined at both a whole-brain and region of interest (ROI) level, with ROIs defined either anatomically or based on clusters derived from the group data.
Cognitive function | Baseline to Day 14
  A standard test battery will be used to examine changes in behavioural measures of cognition, including speed of processing (detection task), attention/vigilance (identification task), working memory, visual learning and memory, and reasoning and problem solving. In addition, a visual analogue scales (VAS) will be used to assess subjective mood state.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for Study 201131 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201131?search=study&study_ids=201131#rs